CLINICAL TRIAL: NCT06730919
Title: Risk Factors for Postpartum Hemorrhage After Cesarean Delivery in Women With Systemic Autoimmune Disease: A Multicenter Retrospective Study
Brief Title: Risk Factors for Postpartum Hemorrhage
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LY2024-274-B
Record Dates: First submitted 2024-12-08; First posted 2024-12-12 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Postpartum Hemorrhage; Systemic Autoimmune Diseases
Keywords: postpartum hemorrhage; systemic autoimmune disease; cesarean delivery; risk factors
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PPH group: The EBL after cesarean delivery within 24 h over 1000mL
  Interventions: Diagnostic Test: Estimated Blood Loss after cesarean delivery within 24 h
- Non-PPH group: The EBL after cesarean delivery within 24 h not over 1000mL

INTERVENTIONS:
Diagnostic Test: Estimated Blood Loss after cesarean delivery within 24 h — The total estimated blood loss was calculated by equation: Estimated Blood Loss (EBL) = EBV ×((HCT1 - HCT2)/(HCT mean)), EBV = Estimated Blood volume; whereas EBV = Patient's weight (in kilogram) × 70 mL/kg, HCT1=preoperative hematocrit, HCT2 = postoperative hematocrit, and HCT mean = (HCT1 + HCT2)/2
  Groups: PPH group

SUMMARY:
Postpartum hemorrhage (PPH) is the most significant leading cause of pregnancy-related mortality in high-risk cesarean delivery women. Systemic autoimmune diseases are associated with adverse pregnancy outcomes (APOs), including PPH, preeclampsia, thromboembolism, abortion, and intrauterine growth restriction. The incidence of PPH in women with systemic lupus erythematosus (SLE) has been reported to be as high as 34%. However, few studies have investigated PPH risk factors in pregnant women with systemic autoimmune disease. Therefore, the purpose of this study is to investigate the incidence and related risk factors of PPH in pregnant women with systemic autoimmune disease, and to provide the latest evidence for further study on prevention of PPH in women at high risk of PPH.

DETAILED DESCRIPTION:
The worldwide estimated cumulative prevalence of autoimmune disease is approximately 5%. Studies are often limited by small sample sizes and focused on a specific autoimmune disease such as SLE and antiphospholipid syndrome (APS), which is characterized by the production of autoantibodies leading to inflammation of multiple organs. Systemic autoimmune diseases are associated with APOs, including increased cesarean delivery rates, PPH, preeclampsia, thromboembolism, abortion, premature delivery, and intrauterine growth restriction. Preeclampsia is the most commonly reported complication in patients with SLE and is also a high risk factor for PPH. The incidence of PPH in women with SLE has been reported to be as high as 34%. Antiphospholipid antibodies (APLAs) are often present in SLE and APS patients, which predict serious perinatal complications and are associated with the risk of thrombosis. APLAs are detected not only in SLE and APS but also in other connective tissue diseases such as systemic sclerosis (SSc), Sjögren's syndrome (SS), rheumatoid arthritis (RA), and undifferentiated connective tissue disease (UCTD). Women with positive APLAs during pregnancy usually receive antithrombotic therapy to reduce the incidence of fetal loss, which may increase the risk of PPH, but existing research evidence is insufficient. PPH increases the need for blood transfusion and related complications and is a significant clinical and socio-economic problem. The aim of this study is to investigate the incidence and related risk factors of PPH in pregnant women with systemic autoimmune disease, and to provide the latest evidence for further study on prevention of PPH in women at high risk of PPH.

The investigators will review patients who underwent cesarean delivery in five hospitals between June 2019 and June 2024. The complication of pregnancy, placental function, estimated blood loss 24h postoperatively, blood transfusion 3d postpartum, additional uterotonics, other surgical intervention for PPH and APOs will be recorded. The group of patients included in the analysis for risk factors associated with PPH consisted of those who with systemic autoimmune disease.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational period was ≥ 28 week;
2. Delivered by cesarean delivery;
3. With systemic autoimmune diseases (SLE, APS, SSc, SS,RA, UCTD)

Exclusion Criteria:

1. Intrauterine fetal death
2. Hemorrhagic disease, significant prenatal bleeding
3. Missing clinical information

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All women with systemic autoimmune diseases who underwent cesarean delivery in Renji Hospital, School of Medicine, Shanghai Jiaotong University, The First Affiliated Hospital, Sun Yat-sen University, Women's hospital school of medicine zhejiang university，Obstetrics & Gynecology Hospital of Fudan University，and Shanghai First Maternity and Infant Hospital between June 2019 and June 2024, and who met the inclusion criteria were eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
The incidence of PPH | From skin incision to 1day after surgery
  PPH is defined as estimated blood loss ≥1000 mL within 24 h after cesarean delivery.

SECONDARY OUTCOMES:
Estimated blood loss within 1day after surgery | From skin incision to 1day after surgery
  Estimated blood loss is calculated by GROSS EQUATION: Estimated Blood Loss (EBL) = EBV ×((HCT1 - HCT2)/(HCT mean)), EBV = Estimated Blood volume; whereas EBV = Patient's weight (in kilogram) × 70 mL/kg, HCT1=preoperative hematocrit, HCT2 = postoperative hematocrit, and HCT mean = (HCT1 + HCT2)/2;
The volume of blood transfusion within 3days after surgery and complications | From skin incision to 3days after surgery
  The volume of blood transfusion within 3days after surgery and complications(such as fever, allergy, hemolysis, renal dysfunction)
Whether additional uterotonics are needed | From the delivery of placenta until 3 days postoperatively.
  Uterotonics other than intraoperative routine dose intravenous and intrauterine infusion of oxytocin.
Whether other surgical intervention for PPH are needed | From the delivery of placenta until 3 days postoperatively.
  Patients who need other surgical intervention(such as intrauterine balloon compression hemostasis, uterine artery ligation or embolization and hysterectomy) to control PPH.
Maternal and neonatal mortality 42d after cesarean delivery | From skin incision to 42 days after surgery.
  All-cause mortality 42d after cesarean delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Xiao, PHD, Study Director — Renji Hospital, Shanghai Jiaotong University, School of Medcine
Locations (5):
- China (5):
  - Renji Hospital, Shanghai Jiaotong University, School of Medcine, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - Women's hospital school of medicine zhejiang university, Hangzhou
  - Obstetrics & Gynecology Hospital of Fudan University, Shanghai
  - Shanghai First Maternity and Infant Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No